CLINICAL TRIAL: NCT06009627
Title: Phase II Clinical Study of Darsilide Combined With Exemestane+Goserelin Neoadjuvant Endocrine Therapy in HR Positive and HER2 Negative Premenopausal Breast Cancer Patients
Brief Title: Study of Neoadjuvant Endocrine Therapy in HR Positive and HER2 Negative Premenopausal Breast Cancer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tianjin Hospital Cancer
Record Dates: First submitted 2023-07-18; First posted 2023-08-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Injections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dalpiciclib+Goserelin+Exemestane (Experimental): SD patients undergoing 2 cycles of preoperative treatment were randomly assigned to Group A and received darcelli, Exemestane, and Goserelin
  Interventions: Drug: dalpiciclib、Exemestane、Gosserine
- Docetaxel, epirubicin hydrochloride, Cyclophosphamide (Active Comparator): SD patients undergoing 2 cycles of preoperative treatment were randomly assigned to Group B and received TAC chemotherapy
  Interventions: Drug: Docetaxel for injection、Epirubicin hydrochloride for injection、Cyclophosphamide for injection

INTERVENTIONS:
Drug: dalpiciclib、Exemestane、Gosserine — dalpiciclib: once a day, 125 mg each time, taken for 3 weeks, stopped for 1 week, 1 for 4 weeks
  Period. It is recommended to take the medication at approximately the same time every day, delivered in warm water, on an empty stomach, at least before taking the medication
  Fasting for 1 hour before and after.
  Exemestane: 25mg, oral, once a day, continuous administration.
  Gosserine: 3.6mg, subcutaneous injection, once every four weeks, continuous administration
  Arms: dalpiciclib+Goserelin+Exemestane
Drug: Docetaxel for injection、Epirubicin hydrochloride for injection、Cyclophosphamide for injection — Docetaxel for injection: 75mg/m2, intravenous drip, approximately 30 minutes. Dose reduction and delayed administration are allowed every three weeks, with a maximum of three weeks of delayed administration allowed since the last administration time
  Calculate, otherwise terminate treatment.
  5. Epirubicin hydrochloride for injection: 75mg/m2, intravenous drip. Once every three weeks, allowing for dose reduction
  And delayed administration, with a maximum allowable delay of 3 weeks, calculated from the last administration time. Otherwise
  Stop treatment.
  6. Cyclophosphamide for injection: 500mg/m2, intravenous drip. Once every three weeks, allowing for dose reduction and
  Delayed administration, allowed up to 3 weeks, calculated from the last administration time, otherwise terminated treat
  Arms: Docetaxel, epirubicin hydrochloride, Cyclophosphamide

SUMMARY:
A multicenter, prospective, open, randomized cohort, non controlled phase II clinical study to evaluate the effectiveness and safety of Darxil combined with Exemestane+goserelin neoadjuvant endocrine therapy in HR positive and HER2 negative premenopausal breast cancer patients. The study object was to evaluate the HR positive and HER2 negative premenopausal breast cancer patients with SD after 2 cycles of neoadjuvant chemotherapy. The main endpoint was the objective response rate (ORR) of treatment

DETAILED DESCRIPTION:
A multicenter, prospective, open, randomized cohort, non controlled phase II clinical study to evaluate the effectiveness and safety of Darxil combined with Exemestane+goserelin neoadjuvant endocrine therapy in HR positive and HER2 negative premenopausal breast cancer patients. The study object was to evaluate the HR positive and HER2 negative premenopausal breast cancer patients with SD after 2 cycles of neoadjuvant chemotherapy. The main endpoint was the objective response rate (ORR) of treatment。Objective: To evaluate the efficacy and safety of darsilide combined with endocrine therapy in SD patients with HR positive and HER2 negative premenopausal breast cancer after 2 cycles of neoadjuvant chemotherapy. It is planned to recruit 119 HR positive and HER2 negative premenopausal breast cancer patients in Group A to conduct the trial with Simon's two-stage design. The null hypothesis is a true response rate of 0.2, while the alternative hypothesis is a true response rate of 0.4. The experiment was conducted in two stages. In the first stage, 13 patients were enrolled. If there are ≤ 3 responses in 13 patients, the study will be stopped Early stopping. Otherwise, continue30 patients were enrolled, with a total sample size of 43. If there are ≥ 13 patients responding, the treatment is effective. Group B was randomly assigned in a 1:1 ratio, with the same number of participants as Group A, resulting in 43 final participants. Calculated based on the proportion of SD patients in 2 cycles of neoadjuvant chemotherapy accounting for 80%, and considering a 10% dropout rate, the final enrollment was made The sample size is 119 cases. The actual samples for molecular testing can be randomly selected based on clinical efficacy, with a statistically significant number.

ELIGIBILITY:
Inclusion Criteria:

* All patients were operable estrogen receptor (ER) positive (>1%), regardless of PR expression level, HER2 receptor negative invasive breast cancer. Follow the 2018 ASCO-CAP HER2 negative interpretation guideline standard. Confirmed by the pathological laboratory that the immunohistochemical (IHC) score is 0 or 1-2+and the in situ hybridization (ISH) test is negative (ISH amplification rate<2.0);
* Stage II-III initial treatment patients whose tumor staging meets the AJCC 8th edition standards;
* At least one measurable breast and/or axillary disease;
* ECOG 0-1, with an estimated lifespan of at least 12 months;
* The functional level of the main organs must meet the following requirements:

Blood routine: ANC ≥ 1.5 × ten9/L; PLT ≥ 90 × ten9/L; Hb ≥ 90 g/L;Blood biochemistry: TBIL ≤ 2.5 × ULN; ALT and AST ≤ 2.5 × ULN; BUN and Cr≤ 1.5 × ULN;

* Lead ECG: QT interval (QTcF) corrected by Fridericia method<470 ms for women;
* Able to accept all puncture biopsies required by the protocol;
* Volunteer to join this study, sign informed consent, have good compliance, and be willing to cooperate with follow-up;
* Women with fertility potential must have a negative Pregnancy test (urine or serum) within 7 days after administration,

And agree to use acceptable birth control methods during the study period to avoid pregnancy.

Exclusion Criteria:

* Received any form of anti-tumor treatment within 28 days prior to the start of the study;
* Simultaneously receiving any anti-tumor treatment beyond the provisions of other protocols;
* Bilateral breast cancer, inflammatory breast cancer or occult breast;
* Stage IV breast cancer;
* Severe dysfunction of important organs such as heart, liver, and kidney;
* Unable to swallow, chronic diarrhea and Bowel obstruction, there are many factors that affect drug taking and absorption;
* Participated in other drug clinical trials within 4 weeks prior to enrollment;
* Those with a known history of allergies to the drug components of this protocol; Have a history of immunodeficiency, including positive Diagnosis of HIV/AIDS test Sex, HCV, active hepatitis B, or other acquired or congenital immunodeficiency diseases Illness or a history of organ transplantation;
* Have ever suffered from any heart disease, including: (1) arrhythmia that requires medication or has clinical significance

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 119 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) for treatment | At the end of the second cycle (each cycle is 21 or 28 days)
  The proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit requirement

SECONDARY OUTCOMES:
Tumor residual load | At the end of the 6 cycle (each cycle is 21 or 28 days)
  The number of cancer cells, tumor size, or total number of cancer lesions in the human body after surgery

OTHER OUTCOMES:
Breast retention rate | At the end of the 6 cycle (each cycle is 21 or 28 days)
  Postoperative breast preservation ratio
Event free lifetime | At the end of the 6 cycle (each cycle is 21 or 28 days)
  The time from the start of randomized clinical trials to the progression of tumors (in any aspect) or death from any cause
Overall survival (OS) | 2years
  Time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: jie 1 ge, 1, Study Director — yes
Locations (1):
- Jie Ge, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No